CLINICAL TRIAL: NCT03810937
Title: Optimal Head and Neck Position for Videolaryngoscopy Intubation
Brief Title: Optimal Head and Neck Position for Videolaryngoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Fahad Specialist Hospital Dammam (Other)
Responsible Party: Principal Investigator, Munir Bamadhaj, Principal Investigator, King Fahad Specialist Hospital Dammam
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ANS004
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Airway Complication of Anesthesia
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in 2 groups:
  * Group sniffing (S): we will start by performing first videolaryngoscopy to find best view in flat position then the anesthesiologist will remove the Glidescope and the patient will be positioned in sniffing position using the pillow and another videolaryngoscopy will be attempted in sniffing position to find best view in this position and the patient will be intubated in this position.
  * Group flat (F): same procedure will be done but starting from sniffing position and the patient will be intubated in flat position.
Who Masked: Participant, Outcomes Assessor
Masking Description: Analysis of the recorded videolaryngoscopic attempts will be performed later by a blinded researcher who was not involved with airway management.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group sniffing (S) (Active Comparator): intervention: Head position changes : we will start by performing first videolaryngoscopy to find best view in flat position then the anesthesiologist will remove the Glidescope and the patient will be positioned in sniffing position using the pillow and another videolaryngoscopy will be attempted in sniffing position to find best view in this position and the patient will be intubated in this position.
  Interventions: Other: head position
- Group Flat (F) (Active Comparator): intervention: Head position changes same procedure will be done but starting from sniffing position and the patient will be intubated in flat position.
  Interventions: Other: head position

INTERVENTIONS:
Other: head position — head positioning in sniffing or flat position

SUMMARY:
The introduction of videolaryngoscopy constituted a revolution in airway management since it could provide better laryngeal exposure (indirect) in situations of difficult or impossible visualization by direct laryngoscopy. The use of Videolaryngoscopes, however, does not always guarantee adequate exposure or end up always in successful tracheal intubation. Failed tracheal intubation with videolaryngoscopy has been reported. We hypothesized that may be the failure was due to omitting some preparatory steps, including optimal head positioning, leading to a less than expected exposure and/or difficult or impossible intubation. There are no recommendations currently from the scientific organizations regarding the optimal head position when using a GlideScope and it is unknown currently whether head position can affect visualization or tracheal intubation attempts when using this device.

DETAILED DESCRIPTION:
* Multicentric,randomized, prospective and controlled study.
* After Institutional Review Board approval, signed written informed consents will be obtained from 165 adult patients with American Society of Anesthesiologists physical status 1-3 who are scheduled for elective surgery requiring endotracheal intubation.
* The following parameters will assessed and documented during the preoperative airway evaluation: BMI, mouth opening, thyromental distance, range of neck movement, and modified Mallampati classification. An 8cm non-compressible pillow.
* Patients will be randomized following coin toss into two groups depending on intubation position; Group Sniffing position(S) for obverse side and group flat position(F) for reverse side
* After premedication, American Society of Anesthesiologists' standard monitors will be applied, and preoxygenation for 3 to 5 minutes will be performed. After anesthesia induction and complete muscle relaxation as evidenced by loss of all evoked adductor pollicis responses to train of four stimulation of the ulnar nerve:
* Group sniffing (S): investigator will start by performing first videolaryngoscopy to find best view in flat position then the anesthesiologist will remove the Glidescope and the patient will be positioned in sniffing position using the pillow and another videolaryngoscopy will be attempted in sniffing position to find best view in this position and the patient will be intubated in this position.
* Group flat (F): same procedure will be done but starting from sniffing position and the patient will be intubated in flat position.
* The laryngoscopist will be asked not to use external laryngeal manipulation and to use the same lifting force throughout the study period. If these maneuvers deemed necessary for tracheal intubation (no visualization of vocal cords from full inflation to full deflation or the reverse, the laryngoscopist will be asked grade the view before applying the maneuver then use the required maneuver and record which intervention was needed and utilized.
* The estimated time to review theses different head elevation degrees is around 45 seconds.
* After preoxygenation technique we have a margin of 6 to 8 minutes of apnea without significant desaturation. Investigator will exclude also patients with high risk of desaturation (obesity and initial low saturation).
* The indirect laryngoscopic views will be graded using the same grading method used for direct laryngoscopy i.e. modified Cormack and Lehane. POGO score (percent of glottis opening viewed) will be also used to subcategorize subjects whose views lie between grade 1 and 3 C&L.

Analysis of the recorded videolaryngoscopic attempts will be performed later by a blinded researcher who was not involved with airway management.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with American Society of Anesthesiologists physical status 1-3 who are scheduled for elective surgery requiring endotracheal intubation.

Exclusion Criteria:

* history of difficult intubation, poor dentition, gastroesophageal reflux disease ,initial low oxygen saturation, severe/morbid obesity (body mass index [BMI] greater than 35 kg/m2),neck deformities, atlano-axial subluxation or at risk of aspiration.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
optimal head position during videolaryngoscopy intubation | intratracheal intubation procedure
  the optimum head position during videolaryngoscopy intubation will be successful first pass tracheal intubation.

SECONDARY OUTCOMES:
best laryngeal exposure | intratracheal intubation procedure
  the best laryngeal exposure (according to modified Cormack and Lehane classification) head position

CONTACTS AND LOCATIONS:
Overall Officials: MUNIR H BAMADHAJ, MD, Principal Investigator — King Fahad Specialist Hospital Dammam
Locations (1):
- King Fahad Specialist Hospital, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No